CLINICAL TRIAL: NCT05151679
Title: Chelated Oral Iron Versus Intravenous Iron Sucrose for Treatment of Iron Deficiency Anemia Late in Pregnancy ( Randomized Controlled Trial )
Brief Title: Chelated Oral Iron Versus Intravenous Iron Sucrose for Treatment of Iron Deficiency Anemia Late in Pregnancy
Status: Available | Type: Expanded Access
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Shaban Mohammed Farghaly, resident doctor, Assiut University
Other Study IDs: oral iron versus I.V iron
Record Dates: First submitted 2021-11-28; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Iron Deficiency Anemia of Pregnancy
MeSH Terms: interventions — Iron Chelating Agents; Ferric Oxide, Saccharated

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Chelated Iron — Treatment will be started 24rh after initial visit women will be randomized used random sequence computer generated list in such a way that every patient had equal chance to be among any of the two groups either to group 1 , where they will receive I.V ferrous sucrose in the E.U in Women's Health Hospital Assuit University as an i.v infusion in 250 ml 0.9% sodium chloride slowly over 30 minutes.
  The total required dose of iron will be divided into three doses, which will be given every 3 days, and the maximum daily dose is 200mg ( 2 ampoules ).
  Other Names: ferrotron
Drug: Iron sucrose — to group 2 where they will receive chelated oral iron, they will be given iron chelated amino acid containing 15 mg of elemental iron once daily for 6 weeks. the women will be advised to take 1 tab of iron chelated amino acid containing 15mg of elemental iron once daily with meals for 6 weeks from the day of recruitment.
  Other Names: sacrofer

SUMMARY:
compare the efficacy and safety of intravenous iron sucrose versus chelated oral iron in the treatment of iron deficiency anemia late in pregnancy.

DETAILED DESCRIPTION:
patients will be recruited from the pregnant women who will attend the outpatient clinic at Women's Health Hospital Assuit University with the diagnosis of iron deficiency anaemia between 26-34 weeks with Hb level 8-10 in the initial visit the patients will be counselled about the iron therapy, its benefits and risk of discontinuation written consent will be obtained.

All women will be subjected to the following:

1. History taking

   1. Personal history: demographic factors, age and dietary habits.
   2. Obstetric history: parity, EDD, last delivery, gestational age determined from last menstrual period or previous early ultrasound scanning report.
   3. Past history: history of chronic diseases such as diabetes or hypertension, blood transfusion and either oral or i.v iron treatment.
2. Clinical examination General examination including pulse, blood pressure, BMI, pallor, temperature and auscultation of lungs and heart.

   Abdominal examination for fundal level. The patients of the study will be randomly divided into two groups Group 1 will be treated by I.V ferrous sucrose Group 2 will be treated by chelated oral iron
3. Invetigations

   * Ultrasonography in the initial visit to assess fetal well being.
   * Blood sample will be taken at recruitment on day 0, day 14, day 28, day 40 of therapy.these time points were chosen on the basis of previous studies and to minimize inconvenience to women.

   The time points were also chosen to detect any difference in the speed of restoration of Hb% and iron stores.

   The blood sample will be examined for the following:
   1. Complete blood picture. A sample of 2 ml venous blood will be collected in EDTA vacutainers.
   2. Serum ferritin evaluation. A sample of 2 ml venous blood will be collected in EDTA vacutainers and separated sera will be stored at 20 C until the time of assay by turbidimetric technique.
   3. Total iron binding capacity. A sample of 2 ml venous blood will be collected in EDTA vacutainers
4. Doses and administration Treatment will be started 24rh after initial visit women will be randomized used random sequence computer generated list in such a way that every patient had equal chance to be among any of the two groups either to group 1 , where they will receive I.V ferrous sucrose in the E.U in Women's Health Hospital Assuit University as an i.v infusion in 250 ml 0.9% sodium chloride slowly over 30 minutes, and then will be discontinued for another 30 minutes to detect any hypersensitivity reactions with monitoring of vital signs during infusion, antishock measures will be prepared beside the patient during administration ( corticosteroids, antihistaminic, calcium and oxygen ). Patients will be asked to note any symptoms or adverse effects of treatment such as facial flushing nausea, metallic taste, dyspepsia, and burning at the site of injection.

The dose in mg will be calculated from the following formula:

2.4 × weight × ( target - actual Hb ) I g/dl + 500 Target Hb 12 g% The total required dose of iron will be divided into three doses, which will be given every 3 days, and the maximum daily dose is 200mg ( 2 ampoules ). This group will not receive further iron supplementation. They will be asked to note any symptoms or adverse effects of treatment.

or to group 2 where they will receive chelated oral iron, they will be given iron chelated amino acid containing 15 mg of elemental iron once daily for 6 weeks. the women will be advised to take 1 tab of iron chelated amino acid containing 15mg of elemental iron once daily with meals for 6 weeks from the day of recruitment. Date will be given when to stop oral supplementation after 6 weeks. This group will be advised to note side effects such as nausea, metallic taste, dyspepsia and constipation.

We will add 500µg of folic acid to patients of group 1 once daily for 6 weeks to eliminate the differences in the results between the groups as ferrotron ( chelated oral iron for second group ) contains 400µg folic acid.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 years or more with established iron deficiency anemia ( Hb: 8-10 )
2. Pregnancy 26-34 weeks

Exclusion Criteria:

1. Anemia due to other causes than iron deficiency anemia.
2. Recent blood transfusion (in the last 3 months ).
3. Allergy to iron.
4. Multiple pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

REFERENCES:
- [Result] Bencaiova G, von Mandach U, Zimmermann R. Iron prophylaxis in pregnancy: intravenous route versus oral route. Eur J Obstet Gynecol Reprod Biol. 2009 Jun;144(2):135-9. doi: 10.1016/j.ejogrb.2009.03.006. Epub 2009 Apr 29. PMID 19406557
- [Result] Means RT. Iron Deficiency and Iron Deficiency Anemia: Implications and Impact in Pregnancy, Fetal Development, and Early Childhood Parameters. Nutrients. 2020 Feb 11;12(2):447. doi: 10.3390/nu12020447. PMID 32053933